CLINICAL TRIAL: NCT00644124
Title: A Phase I Open-label Dose-escalation Study of Intravenous Aflibercept (AVE0005, VEGF Trap) in Combination With R-CHOP Administered Every 2 Weeks or Every 3 Weeks in Patients With Non Hodgkin's B-cell Lymphoma
Brief Title: Aflibercept and Standard Chemotherapy (R-CHOP) in First Line of Non Hodgkin B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD10173; EudraCT 2007-003737-16
Record Dates: First submitted 2008-03-21; First posted 2008-03-26 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin's lymphoma; angiogenesis inhibitors; CHOP protocol
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aflibercept RCHOP 14 (Experimental): Aflibercept (25 mg/ml by IV over an hour) in combination with fixed dose of rituximab (R), cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) administered every 2 weeks. A dose of 2.0 mg/kg administered as Dose Level 1, 4.0 mg/kg as Dose Level 2, and 6.0 mg/kg dose as Dose level 3.
  Interventions: Drug: aflibercept
- Aflibercept RCHOP 21 (Experimental): Aflibercept (25 mg/ml by IV over an hour) in combination with fixed dose of rituximab (R), cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) administered every 3 weeks. A dose of 3.0 mg/kg administered as Dose Level 1, 6.0 mg/kg as Dose Level 2, and 8.0 mg/kg dose as Dose level 3.
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — in combination with standard treatment R-CHOP

SUMMARY:
The purpose of this study is to determine the selected dose of aflibercept when it is combined with R-CHOP treatment (Rituximab/Cyclophosphamide/Doxorubicin/Vincristine/Prednisone +/- intrathecal Methotrexate) administered every 2 weeks or every 3 weeks, in non Hodgkin B-cell lymphoma, and to determine how the body handles aflibercept when it is administered with R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-Hodgkin B-cell lymphoma, good condition, not previously treated

Exclusion Criteria:

* Contraindication to any drug contained in the R-CHOP (Rituximab/Cyclophosphamide/Doxorubicin/Vincristine/Prednisone +/- intrathecal Methotrexate)
* Less than 42 days elapsed from prior major surgery (28 days from other prior surgery) to the time of inclusion
* Cerebral or leptomeningeal involvement.
* History of another neoplasm (Adequately treated basal cell or squamous cell skin cancers, carcinoma in situ of the cervix, or any other cancer from which the patient has been disease free for > 5 years are allowed)
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to the first drug intake
* Any acute or chronic medical condition, which could impair the ability of the patient to participate to the study or could interfere with interpretation of study results
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* Abnormal kidney function
* Evidence of clinically significant bleeding diathesis, non-healing wound or underlying coagulopathy
* Pregnant or breast-feeding woman, or patient with reproductive potential (male, female) without an effective method of contraception
* History of hypersensitivity to any Trap agents or recombinant proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
selected dose of aflibercept based on Dose Limiting Toxicities observed | cycle 1 +/- 2

SECONDARY OUTCOMES:
Adverse events | treatment period
Response rate | cycle 2, 4 and 8
Progression free survival | study period
Biomarkers | Study period

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Haioun, MD, Principal Investigator — Groupe d'Etudes du Lymphome de l'Adulte
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France